CLINICAL TRIAL: NCT06869278
Title: An Open Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of LCAR-AIO CAR-T Cells for Treating Relapsed/Refractory Neurological Autoimmune Diseases
Brief Title: A Study of LCAR-AIO CAR-T Cells for Treating Relapsed/Refractory Neurological Autoimmune Diseases
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Nanjing Legend Biotech Co. (Industry)
Responsible Party: Principal Investigator, Qiubai Li, Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LB2305-0003
Record Dates: First submitted 2025-02-25; First posted 2025-03-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Multiple Sclerosis (MS); Neuromyelitis Optica Spectrum Disease (NMOSD); Anti-Myelin Oligodendrocyte Glycoprotein-IgG Associated Disorders (MOGAD); Myasthenia Gravis
Keywords: Relapsed/Refractory Multiple Sclerosis (r/r MS); Relapsed/Refractory Neuromyelitis Optica Spectrum Disease (r/r NMOSD); Relapsed/Refractory Anti-Myelin Oligodendrocyte Glycoprotein-IgG Associated Disorders (r/r MOGAD); Relapsed/Refractory Myasthenia Gravis (r/r MG)
MeSH Terms: conditions — Multiple Sclerosis; Myasthenia Gravis; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LCAR-AIO T Cells (Experimental): Chimeric antigen receptor T cells (LCAR-AIO) Each subject will be given a single-dose LCAR-AIO cells infusion at each dose level
  Interventions: Biological: LCAR-AIO T cells

INTERVENTIONS:
Biological: LCAR-AIO T cells — Before treatment with LCAR-AIO T cells, subjects will receive a conditioning regimen.

SUMMARY:
This is a prospective, single-arm, open-label, dose-exploration and expansion clinical study of LCAR-AIO in adult subjects with relapsed/refractory neurological autoimmune diseases.

DETAILED DESCRIPTION:
This is a prospective, single-arm, open-label exploratory clinical study to evaluate the safety, tolerability, pharmacokinetics and efficacy profiles of LCAR-AIO, a chimeric antigen receptor (CAR) -T cell therapy in subjects with relapsed/refractory neurological autoimmune diseases. Patients who meet the eligibility criteria will receive LCAR-AIO infusion. The study will include the following sequential stages: screening, apheresis, pre-treatment (cell product preparation: lymphodepleting chemotherapy), treatment (LCAR AIO infusion) and follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participate in clinical research.
2. Age 18-70 years.
3. Adequate organ function at screening.
4. Clinical laboratory values meet criteria at screening visit.
5. Indications include:

MS;

1. Have been diagnosed of MS at least 6 months before screening.
2. Fulfill relapsed/refractory MS conditions.

NMOSD/MOGAD:

1. Have been diagnosed of NMOSD/MOGAD at least 6 months before screening.
2. AQP-4 IgG (NMOSD), or MOG-IgG (MOGAD) should be positive by CBA (Cell based transfection immunofluorescence assay).
3. Fulfill relapsed/refractory NMOSD/MOGAD conditions.

MG:

1. Have been diagnosed of MG at least 6 months before screening.
2. AChR-IgG or MuSK-IgG should be positive.
3. Fulfill relapsed/refractory NMOSD/MOGAD conditions.

Exclusion Criteria:

1. Active infections such as hepatitis and tuberculosis.
2. Other autoimmune diseases.
3. Serious underlying diseases such as tumor, uncontrolled diabetes and clinically significant cardiovascular disease.
4. Female subjects who were pregnant, breastfeeding, or planning to become pregnant while participating in this study or within 1 year of receiving LCAR-AIO treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2025-06-17 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence, severity, and type of treatment-emergent adverse events (TEAEs) | Baseline to 104 Weeks after last subject infusion
  An adverse event refers to any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product (investigational or non-investigational), which does not necessarily have a causal relationship with the treatment.
Incidence of dose-limiting toxicity (DLT) | 30 days after LCAR-AIO infusion (Day 1)
  DLTs are severe adverse events refers to any untoward medical occurred in a subject participated in a clinical investigation, which have a causal relationship with the treatment and will limit the dose escalation.
Chimeric Antigen Receptor T (CAR-T) Positive Cell Concentration | Baseline to 104 Weeks after last subject infusion
  Venous blood samples will be collected for measurement of CAR-T positive cellular concentration.
Recommended Phase 2 Dose (RP2D) regimen finding | Baseline to 104 Weeks after last subject infusion
  RP2D established through dose exploratory.
Transgene Levels of LCAR-AIO CAR-T Cells | Baseline to 104 Weeks after last subject infusion
  Transgene Levels of LCAR-AIO CAR-T Cells using sensitive assay methods will be assessed

SECONDARY OUTCOMES:
Annua Relapse Rate (ARR) | Baseline to 104 Weeks after last subject infusion
  ARR refers to the number of relapses divided by observed year after LCAR-AIO infusion.
Change in Expanded Disability Status Scale (EDSS) scores from baseline up to 104 weeks | Baseline to 104 Weeks after last subject infusion
  The EDSS is a method of quantifying disability and monitoring changes in the level of disability over time. EDSS score ranges from 0 (normal neurological exam) to 10 (death from MS). A negative change from baseline indicates improvement.
Changes in Visual Acuity from baseline up to 104 weeks | Baseline to 104 Weeks after last subject infusion
  The Visual Acuity is determined by Snellen chart and visual field.
Changes in Visual analogue scale (VAS) pain score from baseline up to 104 weeks | Baseline to 104 Weeks after last subject infusion
  VAS pain score is used to evaluate pain. Line from 0 = no pain to10 = worst pain.
Changes in MSE proportion from baseline up to 104 weeks | Baseline to 104 Weeks after last subject infusion
  The proportion of patients who achieve Minimal Symptom Expression (MSE, defined as reaching an MG-ADL=0~1 or QMGS=0~2) after LCAR-AIO infusion.
Changes in Quantitative Myasthenia Gravis Score (QMGS) from baseline up to 104 weeks | Baseline to 104 Weeks after last subject infusion
  The QMGS is a 13-item scale used to quantify disease severity in MG. The scale measures ocular, bulbar, respiratory, and limb function, grading each finding, and ranges from 0 (no myasthenic findings) to 39 (maximal myasthenic deficits).
Changes in Myasthenia Gravis Activities of Daily Living (MG-ADL) score from baseline up to 104 weeks | Baseline to 104 Weeks after last subject infusion
  The MG-ADL is an eight-question survey of symptom severity. The average level of daily activity function in the last 7 days was assessed and the total score was calculated. Each question response graded from 0 (normal) to 3 (most severe). Cumulative MG-ADL scores range from 0 to 24.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The Affiliated Hospital of Fujian Medical University, Fuzhou
  - The First Affiliated Hospital of SOOCHOW University, Suzhou
  - Union Hospital Tongji Medical College HUAZHONG University of Science and Technology, Wuhan

IPD SHARING:
Plan to Share IPD: No